CLINICAL TRIAL: NCT03946228
Title: Reducing Sedentary Behavior to Improve Sleep: an Ancillary Study to the RESET BP Clinical Trial
Acronym: RESET-SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Kline, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY18120122; R01HL147610 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Sleep; Obstructive Sleep Apnea; Insomnia
Keywords: blood pressure; sedentary behavior; physical activity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders; Sedentary Behavior; Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): The intervention will use behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts to target a 2-4 hour/day reduction in sedentary behavior.
  Interventions: Behavioral: Behavioral Intervention
- Control Condition (No Intervention): Participants randomized to the control condition will receive no intervention during the study. After the 3-month assessment, control participants will be provided with a wrist-worn activity monitor and will be offered the 3-month delayed intervention if desired to aid in retention and recruitment.

INTERVENTIONS:
Behavioral: Behavioral Intervention — The intervention will be delivered by trained research staff who are exercise physiologists or behavioral lifestyle counselors. This target reflects a recent expert statement concluding that desk-based workers should reduce workday sedentary behavior by 2-4 hr (by increasing standing and movement). The approach will combine: behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts. The initial in-person session will occur at the participant's office location. During months 2 and 3, one-on-one in-person meetings will occur at the research lab. Telephone intervention contacts will occur in the 3rd week of months 1-3.
  Arms: Behavioral Intervention

SUMMARY:
Using a multi-method sleep assessment approach, the purpose of this study is to examine the bidirectional relationship between sleep and sedentary behavior in the context of a randomized trial investigating the impact of sedentary behavior reduction on blood pressure.

DETAILED DESCRIPTION:
Disturbed sleep, most notably insomnia and obstructive sleep apnea (OSA), is highly prevalent and associated with increased risk for elevated blood pressure (BP) and cardiovascular disease. Unfortunately, despite the substantial public health burden of disturbed sleep, standard treatments are often limited by poor adherence, inadequate availability, and/or significant side effects. As such, identification of alternative approaches to mitigate disturbed sleep is greatly needed. In contrast to increasing engagement in exercise, we propose that reducing sedentary behavior (SED), or time spent sitting, is a novel and feasible approach to reduce sleep disturbance. We also propose that the presence of disturbed sleep during the intervention could blunt the adherence to attempted SED reduction and impact its cardiovascular health benefits. Therefore, the goal of this ancillary study is to test the hypotheses that SED reduction will improve sleep and that the presence of baseline sleep disturbance will reduce the effectiveness of SED reduction efforts. We will test this hypothesis by adding comprehensive sleep assessments to an ongoing randomized clinical trial (NCT03307343) that is examining the effect of SED reduction on BP. In this parent trial, 300 desk workers with elevated BP are randomized to a 3-month multicomponent behavioral intervention aimed at replacing 2-4 hr/day of SED with light-intensity activity or a 3-month no-contact control condition.

Anticipating the ability to enroll 150 participants from the remaining sample of the parent trial (estimated N~210), we will assess sleep at baseline and post-intervention using 7 nights of wrist-worn actigraphy and 1 night of home-based polysomnography (PSG), yielding objective measures of sleep quality (WASO), total sleep time (TST), OSA severity (apnea-hypopnea index [AHI]), and sleep depth (slow-wave sleep [SWS]. These data will allow us to efficiently address the following specific aims:

Aim 1: To evaluate the effect of a 3-month SED reduction intervention on objective measures of sleep quality, depth, duration, and OSA severity.

Hypothesis: Participants randomized to the SED reduction intervention will have greater reduction than control participants in actigraphy-assessed WASO (primary outcome [hypothesis 1.1]), PSG-assessed AHI and SWS, and greater increase in actigraphy-assessed TST (secondary outcomes [hypothesis 1.2]).

Aim 2: To examine the effect of baseline disturbed sleep on SED reduction and BP improvement.

Hypothesis: Intervention-induced reductions in SED (hypothesis 2.1) and BP (hypothesis 2.2) will be smaller among individuals with disturbed sleep (e.g., elevated WASO or AHI) at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65 years
2. SBP of 120-159 mmHg or DBP of 80-99 mmHg
3. Physically inactive or insufficiently active (i.e., not meeting current aerobic MVPA recommendations [≥150 min/wk])
4. Currently perform deskwork for ≥ 20 hr/wk at a desk compatible with a sit-stand desk attachment
5. Employment within 25-mi radius of University of Pittsburgh
6. Stable employment (≥ 3 mo at current job, plan to be in current job for at least the next 3 mo)
7. Supervisor approval to join intervention
8. Possession of cellular phone able to receive text messages

Exclusion Criteria:

1. SBP ≥ 160 mmHg or DBP ≥ 100 mmHg
2. Use of anti-hypertensive or glucose-controlling medication
3. Comorbid condition that would limit ability to reduce sedentary behavior (e.g., musculoskeletal condition)
4. History of ischemic heart disease, chronic heart failure, stroke, or chronic kidney disease
5. Inability to obtain consent from primary care provider/physician to participate
6. Current use of a sit-stand desk or sedentary behavior prompting device
7. Current enrollment in a weight loss or exercise program, recent (< 1 yr) or planned bariatric surgery
8. Plans to be away from work for an extended period (>1 wk) during the study period
9. Current or recent (within last 6 mo) pregnancy; current or recent (within last 3 mo) breastfeeding
10. Undiagnosed severe OSA (AHI ≥ 30) or insomnia (ISI ≥ 22)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline actigraphic wake after sleep onset (WASO) at 3 months | 3 months
  Primary outcome for Aim 1: actigraphy-assessed wake after sleep onset, averaged over 7 nights
Change from baseline activPAL-assessed sedentary behavior (SED) at 3 months | 3 months
  Primary outcome for Aim 2: SED, assessed via activPAL inclinometer, averaged over 7 days
Change from baseline resting systolic blood pressure (SBP) at 3 months | 3 months
  Primary outcome for Aim 2: resting SBP, measured via oscillometric device following a 10-minute rest averaged over two separate occasions

SECONDARY OUTCOMES:
Change from baseline total sleep time (TST) at 3 months | 3 months
  Secondary outcome for Aim 1: actigraphy-assessed TST, averaged over 7 nights
Change from baseline apnea-hypopnea index (AHI) at 3 months | 3 months
  Secondary outcome for Aim 1: polysomnography-assessed AHI, assessed over 1 night of home-based recording
Change from baseline slow-wave sleep (SWS) at 3 months | 3 months
  Secondary outcome for Aim 1: polysomnography-assessed slow-wave sleep, assessed over 1 night of home-based recording
Change from baseline 24-hour blood pressure at 3 months | 3 months
  Secondary outcome for Aim 2: blood pressure, assessed by an ambulatory monitor during a workday and overnight for 24 hours total
Change from baseline pulse wave velocity (PWV) at 3 months | 3 months
  Secondary outcome for Aim 2: carotid-femoral and carotid-radial PWV, assessed via tonometry following a 10-minute rest

OTHER OUTCOMES:
Change from baseline self-reported sleep patterns at 3 months | 3 months
  Self-reported sleep patterns will be assessed via a daily diary; mean and measures of variability will be obtained from 7 nights of data
Change from baseline Epworth Sleepiness Scale (ESS) scores at 3 months | 3 months
  The ESS, a measure of daytime sleepiness, will be administered at baseline and 3 months; total score will be used
Change from baseline Insomnia Severity Index (ISI) scores at 3 months | 3 months
  The ISI, a measure of insomnia symptom severity, will be administered at baseline and 3 months; total score will be used
Change from baseline Functional Outcomes of Sleep Questionnaire (FOSQ) scores at 3 months | 3 months
  The 10-item version of the FOSQ, a measure of daytime dysfunction due to poor sleep, will be administered at baseline and 3 months; total score will be used
Change from baseline PROMIS Sleep-related Impairment scale scores at 3 months | 3 months
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep-related Impairment Scale, a measure of daytime impairment, will be administered at baseline and 3 months; total score will be used
Change from baseline Pittsburgh Sleep Quality Index (PSQI) scores at 3 months | 3 months
  PSQI will be administered at baseline and 3 months; global score and 3 factors (sleep efficiency, perceived sleep quality, daily disturbances) will be used
Change from baseline actigraphic sleep patterns at 3 months | 3 months
  Actigraphic sleep patterns will be assessed with the Actiwatch Spectrum Plus; mean and measures of variability will be obtained from 7 nights of data
Change from baseline polysomnography (PSG)-assessed sleep patterns at 3 months | 3 months
  Polysomnography will be performed in the participant's home at baseline and 3 months
Change from baseline weight at 3 months | 3 months
  Weight will be measured by digital scale at baseline and 3 months
Change from baseline glucose at 3 months | 3 months
  Glucose will be measured from a fasting blood draw at baseline and 3 months
Change from baseline insulin at 3 months | 3 months
  Insulin will be measured from a fasting blood draw at baseline and 3 months
Change from baseline accelerometer-assessed physical activity at 3 months | 3 months
  Physical activity will be assessed via waist-worn ActiGraph GT3X accelerometer at baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Kline, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Pittsburgh Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified data that are relevant to the primary aims of the study will be provided to external investigators along with a relevant data dictionary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year following peer-reviewed publication of research questions outlined in grant and ending 5 years following publication of study results
Access Criteria: Data access will be provided to external researchers who provide a methodologically sound proposal for secondary data analysis that is approved by the investigators of the study. Proposals should be directed to the study PI.

DOCUMENTS (1):
  • Informed Consent Form (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT03946228/ICF_000.pdf